CLINICAL TRIAL: NCT05974748
Title: Comparative Evaluation of Propolis and Sodium Hypochlorite as Endodontic Irrigants on Post-Operative Pain in Patients With Symptomatic Irreversible Pulpitis
Brief Title: Role of Propolis Endodontic Irrigant on Post-Operative Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Tayyaba Tahira, Lecturer, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2908
Record Dates: First submitted 2023-07-16; First posted 2023-08-03 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Post-operative Pain; Symptomatic Irreversible Pulpitis
Keywords: Propolis; Endodontic Irrigant
MeSH Terms: conditions — Pain, Postoperative | interventions — Propolis

STUDY DESIGN:
Intervention Model Description: 2 interventional groups assigned. 1 will be receiving routine intervention and other is the experimental group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be aware of their interventional group. A proforma and pain intensity scale will be provided to the patient by an intern not involved in the study, to be completed at 24, 48, and 72 hours following the procedure to assess post-operative pain. this proforma will be collected and assessed by the intern.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Hypochlorite (Active Comparator): 5.25% sodium hypochlorite is the gold standard endodontic irrigant. Other Name: NaOCl
  Interventions: Drug: Sodium hypochlorite 5.25%
- Propolis (Experimental): Hydroalcoholic 20% propolis will be used as an endodontic irrigant. Other Name: Bee glue
  Interventions: Drug: Propolis 20%

INTERVENTIONS:
Drug: Sodium hypochlorite 5.25% — The participants will be randomly divided into two groups using the sealed envelope method during the instrumentation process. The clinician will use the irrigation in accordance with the protocol. Between each instrument in group A, 3 ml of 5.25% sodium hypochlorite (NaOCl) will be used to irrigate each canal.
  Other Names: NaOCl
  Arms: Sodium Hypochlorite
Drug: Propolis 20% — In group B, a 20% hydroalcoholic propolis solution of 3 milliliters will be used to irrigate each canal, between each instrument.
  Other Names: Bee glue
  Arms: Propolis

SUMMARY:
The goal of this clinical trial is to compare propolis and sodium hypochlorite as endodontic irrigants in patients presenting with symptomatic irreversible pulpitis.

. The main question it aims to answer is:

• if there is any analgesic effects of 20% Propolis compared with 5.25% NaOCl on the intensity of post-operative pain in patients with symptomatic irreversible pulpitis using VAS pain score. Participants will undergo root canal treatment of their teeth using either 20% propolis solution or 5.25% NaOCl in their first visit of a multi-visit root canal treatment.

Researchers will compare 20% Propolis and 5.25% NaOCl to see reduction in Intensity of Post-Operative Pain using visual analogue scale over 72 hour duration.

DETAILED DESCRIPTION:
Sodium hypochlorite as an endodontic irrigant, poses problems of toxicity. Additionally, its unfavorable odor, taste, failure to remove the smear layer, and proteolytic effect have deleterious effects on the dentine, creating unfavorable structural and mechanical alterations . To get beyond NaOCl limits and adverse effects, it is necessary to look for a biocompatible, equally effective, and dentine friendly irrigant with greater patient acceptance in taste and odor.

The literature lacks an in-vivo study that investigates the anti-inflammatory with analgesic characteristics of Propolis on post-endodontic pain as an irrigant, in patients with symptomatic irreversible pulpitis. This research will endeavor to fill this gap in literature.

ELIGIBILITY:
Inclusion Criteria:

1. ASA-I and II individuals who are between the ages of 18 and 60 years.
2. Patients with mandibular and maxillary premolars who have been diagnosed with symptomatic irreversible pulpitis (with either a normal periapex or symptomatic apical periodontitis).
3. Patients who score moderate to severe (4-10) on a preoperative visual analogue scale (VAS=1-10)

Exclusion Criteria:

1. Patients suffering from severe pain because of traumatic occlusion.
2. Teeth with extensive damage, calcified canals, periapical radiolucency, root resorption, and an open apex.
3. Patients with compromised medical condition (ASA-III and above)
4. Patients who are unable to communicate effectively in either Urdu or English.
5. Pregnant and lactating ladies
6. Patients who are allergic to honey or bee pollen.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Change in post-operative pain intensity on visual analogue scale(0-10) | 24 hours, 48 hours and 72 hours
  Self recorded by patient and then assessed by an intern on a visual analogue scale of 0-10 with 0 being no pain , 10 being worst pain

SECONDARY OUTCOMES:
Need of rescue medicine in both groups | within first 24 hours
  Self recorded by patient and then assessed by an intern on a visual analogue scale of 0-10 with 0 being no pain , 10 being worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Tayyaba Tahira, BDS FCPS, Principal Investigator — Dow International Dental College, Dow University of Health Sciences; Farah Naz, BDS FCPS, Study Director — Dow International Dental College, Dow University of Health Sciences
Locations (1):
- Dow International Dental College, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Only investigators and co-investigators of this study will be able to access to participants' personal data.
  Ownership of the data will remain with the principal investigator and Department of Operative Dentistry, Dow International Dental College(DIDC) , Dow University of Health Sciences